CLINICAL TRIAL: NCT02942667
Title: Magnetic Resonance Imaging of Human Biometrics
Acronym: MRI HB
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: MRI HB
Record Dates: First submitted 2016-09-30; First posted 2016-10-24 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Volunteers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects undergoing high quality MRI Scans

SUMMARY:
The primary objective is to collect high quality MRI data (un-processed or processed) from participating subjects for Medtronic research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age
* Subject is willing and able to undergo study requirements

Exclusion Criteria:

* Subject has a medical condition that precludes the subject from participation
* Subject has any magnetizable foreign object (e.g. jewelry) which cannot be removed for the duration of the study
* Subject is claustrophobic
* Subject is unable to stand without assistance
* Subject requires sedation for MRI scans
* Subject is implanted with non-Magnetic Resonance conditional or other medical device:

  * Non-MRI conditional pacemaker, Implantable Cardiac Defibrillator (ICD), Cardiac Resynchronization Therapy (CRT), or an implantable hemodynamic monitor
  * Metal clips (i.e. brain aneurysm clip)
  * Artificial heart valve
  * Implanted neural stimulator
  * Gastric capsule camera
  * Swan Ganz catheter
  * Stent
  * Inferior Vena Cava (IVC) filter
  * Orthopedic implant
  * Eye prosthesis
  * Vascular access port
  * Penile prosthesis
  * Intrauterine device
* Subject has a cochlear implant, middle ear prosthesis, or has had ear surgery
* Subject has ocular foreign bodies (i.e. metal shavings)
* Subject has any type of device held in place by a magnet (i.e. dentures)
* Subject has an insulin pump
* Subject has metal shrapnel
* Subject is pregnant or lactating
* Subject has magnetizable implant
* Subject requires legally authorized representative to sign Patient Informed Consent (PIC)/ Informed Consent (IC) form
* Subject has other contraindication for an MRI scan as defined by the study site

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll up to 30 subjects at up to 5 study sites in the US.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Collect High Quality MRI Data | Approximately 6 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No